CLINICAL TRIAL: NCT00005313
Title: Human Lipoprotein Pathophysiology - Subproject: Genetics of Familial Combined Hyperlipidemia
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, John Brunzell, Professor Emeritus, Active, Medicine/Division of Metabolism, University of Washington
Other Study IDs: 10927-B; P01HL030086 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia; Hyperlipidemia, Familial Combined
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia; Hyperlipidemia, Familial Combined

STUDY DESIGN:
Observational Model: Family Based
Oversight: Data Monitoring Committee: No

SUMMARY:
To conduct focused studies of lipoprotein physiology and pathophysiology in genetically characterized patients with the objectives of understanding disease mechanisms, developing better treatments, and identifying and preventing early vascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

Premature vascular disease in young hyperlipidemic subjects remains a major unsolved health problem in terms of pathogenesis and treatment. Research advances have led to new markers for genetic analysis, new methods for studying lipoprotein metabolism and atherosclerotic disease progression and regression, and reference values for diagnosing hyperlipidemia.

DESIGN NARRATIVE:

Attention is focused on the molecular, genetic and pathophysiological basis of the inherited dyslipoproteinemias associated with premature coronary artery disease with particular reference to familial combined hyperlipidemia, familial moderate hypercholesterolemia, familial elevation of Lp(a) and the carrier state for homocysteinemia. Coordinated studies of characterization of the pathophysiological state, the identification of possible molecular biological defects and the evaluation of these results in families by statistical genetic techniques are performed in each disorder. The role of protein mediated intravascular modification of lipoproteins and the role of oxidation of lipoproteins in each disorder will lead to characterization of these genetic lipoprotein abnormalities. The study is a subproject within a program project grant.

The subproject on the genetics of familial combined hyperlipidemia (FCHL) was renewed in 1999 through 2010 to continue mapping the apoB elevating gene l(BEL) level using a genomic search in pedigrees with familial combined hyperlipidemia. The major focus of the genetic analyses are the 15 FCHL families under the BEL segregation analysis model in a power analysis. These families also show the most evidence for segregation at an apoB elevating gene locus. Genotyping for a 10 centimorgan genomic scan has been completed for these families.

ELIGIBILITY:
All participants related to a patient with familial combined hyperlipidemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relatives of patients with familial combined hyperlipidemia
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2001-04; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
No outcome measures for this research | 1980-2003
  Analysis of Familial Data

CONTACTS AND LOCATIONS:
Overall Officials: John Brunzell, Principal Investigator — University of Washington

REFERENCES:
- [Background] Brunzell JD. Are all obese patients at risk for cardiovascular disease? Int J Obes. 1984;8(5):571-8. No abstract available. PMID 6394526
- [Background] Brunzell JD, Sniderman AD, Albers JJ, Kwiterovich PO Jr. Apoproteins B and A-I and coronary artery disease in humans. Arteriosclerosis. 1984 Mar-Apr;4(2):79-83. doi: 10.1161/01.atv.4.2.79. No abstract available. PMID 6422918
- [Background] Iverius PH, Brunzell JD. Human adipose tissue lipoprotein lipase: changes with feeding and relation to postheparin plasma enzyme. Am J Physiol. 1985 Jul;249(1 Pt 1):E107-14. doi: 10.1152/ajpendo.1985.249.1.E107. PMID 4014455
- [Background] Iverius PH, Brunzell JD. Chylomicronemia induced by cimetidine. Gastroenterology. 1985 Sep;89(3):664-6. doi: 10.1016/0016-5085(85)90466-4. PMID 4018506
- [Background] Iverius PH, Brunzell JD. Obesity and common genetic metabolic disorders. Ann Intern Med. 1985 Dec;103(6 ( Pt 2)):1050-1. doi: 10.7326/0003-4819-103-6-1050. PMID 4062124
- [Background] Foster DM, Chait A, Albers JJ, Failor RA, Harris C, Brunzell JD. Evidence for kinetic heterogeneity among human low density lipoproteins. Metabolism. 1986 Aug;35(8):685-96. doi: 10.1016/0026-0495(86)90235-0. PMID 3736409
- [Background] Chait A, Foster DM, Albers JJ, Failor RA, Brunzell JD. Low density lipoprotein metabolism in familial combined hyperlipidemia and familial hypercholesterolemia: kinetic analysis using an integrated model. Metabolism. 1986 Aug;35(8):697-704. doi: 10.1016/0026-0495(86)90236-2. PMID 3736410
- [Background] Angelin B, Hershon KS, Brunzell JD. Bile acid metabolism in hereditary forms of hypertriglyceridemia: evidence for an increased synthesis rate in monogenic familial hypertriglyceridemia. Proc Natl Acad Sci U S A. 1987 Aug;84(15):5434-8. doi: 10.1073/pnas.84.15.5434. PMID 3474660
- [Background] Auwerx JH, Deeb S, Brunzell JD, Peng R, Chait A. Transcriptional activation of the lipoprotein lipase and apolipoprotein E genes accompanies differentiation in some human macrophage-like cell lines. Biochemistry. 1988 Apr 19;27(8):2651-5. doi: 10.1021/bi00408a003. PMID 3401441
- [Background] Iverius PH, Brunzell JD. Relationship between lipoprotein lipase activity and plasma sex steroid level in obese women. J Clin Invest. 1988 Sep;82(3):1106-12. doi: 10.1172/JCI113667. PMID 3417867
- [Background] White JR, Chait A, Klebanoff SJ, Deeb S, Brunzell JD. Bacterial lipopolysaccharide reduces macrophage lipoprotein lipase levels: an effect that is independent of tumor necrosis factor. J Lipid Res. 1988 Oct;29(10):1379-85. PMID 3235920
- [Background] Auwerx JH, Marzetta CA, Hokanson JE, Brunzell JD. Large buoyant LDL-like particles in hepatic lipase deficiency. Arteriosclerosis. 1989 May-Jun;9(3):319-25. doi: 10.1161/01.atv.9.3.319. PMID 2719594
- [Background] Babirak SP, Iverius PH, Fujimoto WY, Brunzell JD. Detection and characterization of the heterozygote state for lipoprotein lipase deficiency. Arteriosclerosis. 1989 May-Jun;9(3):326-34. doi: 10.1161/01.atv.9.3.326. PMID 2719595
- [Background] Auwerx JH, Deeb S, Brunzell JD, Wolfbauer G, Chait A. Lipoprotein lipase gene expression in THP-1 cells. Biochemistry. 1989 May 30;28(11):4563-7. doi: 10.1021/bi00437a009. PMID 2765502
- [Background] Marzetta CA, Foster DM, Brunzell JD. Relationships between LDL density and kinetic heterogeneity in subjects with normolipidemia and familial combined hyperlipidemia using density gradient ultracentrifugation. J Lipid Res. 1989 Sep;30(9):1307-17. PMID 2600538
- [Background] Auwerx JH, Babirak SP, Fujimoto WY, Iverius PH, Brunzell JD. Defective enzyme protein in lipoprotein lipase deficiency. Eur J Clin Invest. 1989 Oct;19(5):433-7. doi: 10.1111/j.1365-2362.1989.tb00255.x. PMID 2511019
- [Background] Langlois S, Deeb S, Brunzell JD, Kastelein JJ, Hayden MR. A major insertion accounts for a significant proportion of mutations underlying human lipoprotein lipase deficiency. Proc Natl Acad Sci U S A. 1989 Feb;86(3):948-52. doi: 10.1073/pnas.86.3.948. PMID 2536938
- [Background] Rohlfing JJ, Brunzell JD. The effects of diuretics and adrenergic-blocking agents on plasma lipids. West J Med. 1986 Aug;145(2):210-8. PMID 2876554
- [Background] Deeb S, Failor A, Brown BG, Brunzell JD, Albers JJ, Motulsky AG. Molecular genetics of apolipoproteins and coronary heart disease. Cold Spring Harb Symp Quant Biol. 1986;51 Pt 1:403-9. doi: 10.1101/sqb.1986.051.01.048. PMID 2884066
- [Background] Weigle DS, Sande KJ, Iverius PH, Monsen ER, Brunzell JD. Weight loss leads to a marked decrease in nonresting energy expenditure in ambulatory human subjects. Metabolism. 1988 Oct;37(10):930-6. doi: 10.1016/0026-0495(88)90149-7. PMID 3173112
- [Background] Austin MA, Brunzell JD, Fitch WL, Krauss RM. Inheritance of low density lipoprotein subclass patterns in familial combined hyperlipidemia. Arteriosclerosis. 1990 Jul-Aug;10(4):520-30. doi: 10.1161/01.atv.10.4.520. PMID 2369363
- [Background] Marzetta CA, Foster DM, Brunzell JD. Conversion of plasma VLDL and IDL precursors into various LDL subpopulations using density gradient ultracentrifugation. J Lipid Res. 1990 Jun;31(6):975-84. PMID 2373965
- [Background] Brunzell JD, Austin MA. Individuality, hyperlipidemia, and premature coronary artery disease. World Rev Nutr Diet. 1990;63:72-83. doi: 10.1159/000418499. No abstract available. PMID 2197808
- [Background] Auwerx JH, Babirak SP, Hokanson JE, Stahnke G, Will H, Deeb SS, Brunzell JD. Coexistence of abnormalities of hepatic lipase and lipoprotein lipase in a large family. Am J Hum Genet. 1990 Mar;46(3):470-7. PMID 1968704
- [Background] Austin MA, Wijsman E, Guo SW, Krauss RM, Brunzell JD, Deeb S. Lack of evidence for linkage between low-density lipoprotein subclass phenotypes and the apolipoprotein B locus in familial combined hyperlipidemia. Genet Epidemiol. 1991;8(5):287-97. doi: 10.1002/gepi.1370080502. PMID 1761202
- [Background] Bruin T, Kastelein JJ, Van Diermen DE, Ma Y, Henderson HE, Stuyt PM, Stalenhoef AF, Sturk A, Brunzell JD, Hayden MR. A missense mutation Pro157 Arg in lipoprotein lipase (LPLNijmegen) resulting in loss of catalytic activity. Eur J Biochem. 1992 Sep 1;208(2):267-72. doi: 10.1111/j.1432-1033.1992.tb17182.x. PMID 1521525
- [Background] Reina M, Brunzell JD, Deeb SS. Molecular basis of familial chylomicronemia: mutations in the lipoprotein lipase and apolipoprotein C-II genes. J Lipid Res. 1992 Dec;33(12):1823-32. PMID 1479292
- [Background] Deeb SS, Failor RA, Brown BG, Brunzell JD, Albers JJ, Motulsky AG, Wijsman E. Association of apolipoprotein B gene variants with plasma apoB and low density lipoprotein (LDL) cholesterol levels. Hum Genet. 1992 Feb;88(4):463-70. doi: 10.1007/BF00215683. PMID 1346774
- [Background] Emmerich J, Beg OU, Peterson J, Previato L, Brunzell JD, Brewer HB Jr, Santamarina-Fojo S. Human lipoprotein lipase. Analysis of the catalytic triad by site-directed mutagenesis of Ser-132, Asp-156, and His-241. J Biol Chem. 1992 Feb 25;267(6):4161-5. PMID 1371284
- [Background] Devlin RH, Deeb S, Brunzell J, Hayden MR. Partial gene duplication involving exon-Alu interchange results in lipoprotein lipase deficiency. Am J Hum Genet. 1990 Jan;46(1):112-9. PMID 2294743
- [Background] Zambon A, Austin MA, Brown BG, Hokanson JE, Brunzell JD. Effect of hepatic lipase on LDL in normal men and those with coronary artery disease. Arterioscler Thromb. 1993 Feb;13(2):147-53. doi: 10.1161/01.atv.13.2.147. PMID 8427851
- [Background] Joven J, Vilella E, Ahmad S, Cheung MC, Brunzell JD. Lipoprotein heterogeneity in end-stage renal disease. Kidney Int. 1993 Feb;43(2):410-8. doi: 10.1038/ki.1993.60. PMID 8441237
- [Background] Hokanson JE, Austin MA, Zambon A, Brunzell JD. Plasma triglyceride and LDL heterogeneity in familial combined hyperlipidemia. Arterioscler Thromb. 1993 Mar;13(3):427-34. doi: 10.1161/01.atv.13.3.427. PMID 8443147
- [Background] Zambon A, Hashimoto SI, Brunzell JD. Analysis of techniques to obtain plasma for measurement of levels of free fatty acids. J Lipid Res. 1993 Jun;34(6):1021-8. PMID 8354949
- [Background] Jarvik GP, Wijsman E, Little RE, Albers JJ, Motulsky AG, Brunzell JD. Host and environmental effects on plasma apolipoprotein B. Int J Clin Lab Res. 1993;23(4):215-20. doi: 10.1007/BF02592312. PMID 8123878
- [Background] Zambon A, Torres A, Bijvoet S, Gagne C, Moorjani S, Lupien PJ, Hayden MR, Brunzell JD. Prevention of raised low-density lipoprotein cholesterol in a patient with familial hypercholesterolaemia and lipoprotein lipase deficiency. Lancet. 1993 May 1;341(8853):1119-21. doi: 10.1016/0140-6736(93)93129-o. PMID 8097805
- [Background] Nevin DN, Brunzell JD, Deeb SS. The LPL gene in individuals with familial combined hyperlipidemia and decreased LPL activity. Arterioscler Thromb. 1994 Jun;14(6):869-73. doi: 10.1161/01.atv.14.6.869. PMID 8199176
- [Background] Jarvik GP, Brunzell JD, Austin MA, Krauss RM, Motulsky AG, Wijsman E. Genetic predictors of FCHL in four large pedigrees. Influence of ApoB level major locus predicted genotype and LDL subclass phenotype. Arterioscler Thromb. 1994 Nov;14(11):1687-94. doi: 10.1161/01.atv.14.11.1687. PMID 7947591
- [Background] Austin MA, Hokanson JE, Brunzell JD. Characterization of low-density lipoprotein subclasses: methodologic approaches and clinical relevance. Curr Opin Lipidol. 1994 Dec;5(6):395-403. doi: 10.1097/00041433-199412000-00002. PMID 7712044
- [Background] Hokanson JE, Krauss RM, Albers JJ, Austin MA, Brunzell JD. LDL physical and chemical properties in familial combined hyperlipidemia. Arterioscler Thromb Vasc Biol. 1995 Apr;15(4):452-9. doi: 10.1161/01.atv.15.4.452. PMID 7749856
- [Background] Yang WS, Nevin DN, Peng R, Brunzell JD, Deeb SS. A mutation in the promoter of the lipoprotein lipase (LPL) gene in a patient with familial combined hyperlipidemia and low LPL activity. Proc Natl Acad Sci U S A. 1995 May 9;92(10):4462-6. doi: 10.1073/pnas.92.10.4462. PMID 7753827
- [Background] Deeb SS, Nevin DN, Iwasaki L, Brunzell JD. Two novel apolipoprotein A-IV variants in individuals with familial combined hyperlipidemia and diminished levels of lipoprotein lipase activity. Hum Mutat. 1996;8(4):319-25. doi: 10.1002/(SICI)1098-1004(1996)8:43.0.CO;2-2. PMID 8956036
- [Background] Yang WS, Nevin DN, Iwasaki L, Peng R, Brown BG, Brunzell JD, Deeb SS. Regulatory mutations in the human lipoprotein lipase gene in patients with familial combined hyperlipidemia and coronary artery disease. J Lipid Res. 1996 Dec;37(12):2627-37. PMID 9017514
- [Background] Wijsman EM, Brunzell JD, Jarvik GP, Austin MA, Motulsky AG, Deeb SS. Evidence against linkage of familial combined hyperlipidemia to the apolipoprotein AI-CIII-AIV gene complex. Arterioscler Thromb Vasc Biol. 1998 Feb;18(2):215-26. doi: 10.1161/01.atv.18.2.215. PMID 9484986
- [Background] Brown BG, Zambon A, Poulin D, Rocha A, Maher VM, Davis JW, Albers JJ, Brunzell JD. Use of niacin, statins, and resins in patients with combined hyperlipidemia. Am J Cardiol. 1998 Feb 26;81(4A):52B-59B. PMID 9526815
- [Background] Carr MC, Hokanson JE, Deeb SS, Purnell JQ, Mitchell ES, Brunzell JD. A hepatic lipase gene promoter polymorphism attenuates the increase in hepatic lipase activity with increasing intra-abdominal fat in women. Arterioscler Thromb Vasc Biol. 1999 Nov;19(11):2701-7. doi: 10.1161/01.atv.19.11.2701. PMID 10559014
- [Background] Ullrich NF, Purnell JQ, Brunzell JD. Adipose tissue fatty acid composition in humans with lipoprotein lipase deficiency. J Investig Med. 2001 May;49(3):273-5. PMID 11352185
- [Background] Purnell JQ, Kahn SE, Schwartz RS, Brunzell JD. Relationship of insulin sensitivity and ApoB levels to intra-abdominal fat in subjects with familial combined hyperlipidemia. Arterioscler Thromb Vasc Biol. 2001 Apr;21(4):567-72. doi: 10.1161/01.atv.21.4.567. PMID 11304474
- [Background] Zambon A, Brown BG, Deeb SS, Brunzell JD. Hepatic lipase as a focal point for the development and treatment of coronary artery disease. J Investig Med. 2001 Jan;49(1):112-8. doi: 10.2310/6650.2001.34107. PMID 11217140
- [Background] Zambon A, Deeb SS, Brown BG, Hokanson JE, Brunzell JD. Common hepatic lipase gene promoter variant determines clinical response to intensive lipid-lowering treatment. Circulation. 2001 Feb 13;103(6):792-8. doi: 10.1161/01.cir.103.6.792. PMID 11171785
- [Background] Carr MC, Kim KH, Zambon A, Mitchell ES, Woods NF, Casazza CP, Purnell JQ, Hokanson JE, Brunzell JD, Schwartz RS. Changes in LDL density across the menopausal transition. J Investig Med. 2000 Jul;48(4):245-50. PMID 10916282
- [Background] Purnell JQ, Kahn SE, Albers JJ, Nevin DN, Brunzell JD, Schwartz RS. Effect of weight loss with reduction of intra-abdominal fat on lipid metabolism in older men. J Clin Endocrinol Metab. 2000 Mar;85(3):977-82. doi: 10.1210/jcem.85.3.6402. PMID 10720026
- [Background] Purnell JQ, Zambon A, Knopp RH, Pizzuti DJ, Achari R, Leonard JM, Locke C, Brunzell JD. Effect of ritonavir on lipids and post-heparin lipase activities in normal subjects. AIDS. 2000 Jan 7;14(1):51-7. doi: 10.1097/00002030-200001070-00006. PMID 10714567
- [Background] Murdoch SJ, Carr MC, Hokanson JE, Brunzell JD, Albers JJ. PLTP activity in premenopausal women. Relationship with lipoprotein lipase, HDL, LDL, body fat, and insulin resistance. J Lipid Res. 2000 Feb;41(2):237-44. PMID 10681407
- [Background] Zambon A, Deeb SS, Bensadoun A, Foster KE, Brunzell JD. In vivo evidence of a role for hepatic lipase in human apoB-containing lipoprotein metabolism, independent of its lipolytic activity. J Lipid Res. 2000 Dec;41(12):2094-9. PMID 11108744
- [Background] Brunzell JD, Hokanson JE. Low-density and high-density lipoprotein subspecies and risk for premature coronary artery disease. Am J Med. 1999 Aug 23;107(2A):16S-18S. doi: 10.1016/s0002-9343(99)00139-4. No abstract available. PMID 10484232
- [Background] Zambon A, Hokanson JE, Brown BG, Brunzell JD. Evidence for a new pathophysiological mechanism for coronary artery disease regression: hepatic lipase-mediated changes in LDL density. Circulation. 1999 Apr 20;99(15):1959-64. doi: 10.1161/01.cir.99.15.1959. PMID 10208998
- [Background] Brunzell JD, Hokanson JE. Dyslipidemia of central obesity and insulin resistance. Diabetes Care. 1999 Apr;22 Suppl 3:C10-3. No abstract available. PMID 10189557
- [Background] Hokanson JE, Brunzell JD, Jarvik GP, Wijsman EM, Austin MA. Linkage of low-density lipoprotein size to the lipoprotein lipase gene in heterozygous lipoprotein lipase deficiency. Am J Hum Genet. 1999 Feb;64(2):608-18. doi: 10.1086/302234. PMID 9973300
- [Background] Franz MJ, Bantle JP, Beebe CA, Brunzell JD, Chiasson JL, Garg A, Holzmeister LA, Hoogwerf B, Mayer-Davis E, Mooradian AD, Purnell JQ, Wheeler M. Evidence-based nutrition principles and recommendations for the treatment and prevention of diabetes and related complications. Diabetes Care. 2002 Jan;25(1):148-98. doi: 10.2337/diacare.25.1.148. No abstract available. PMID 11772915
- [Background] Love MW, Craddock AL, Angelin B, Brunzell JD, Duane WC, Dawson PA. Analysis of the ileal bile acid transporter gene, SLC10A2, in subjects with familial hypertriglyceridemia. Arterioscler Thromb Vasc Biol. 2001 Dec;21(12):2039-45. doi: 10.1161/hq1201.100262. PMID 11742882
- [Background] McNeely MJ, Edwards KL, Marcovina SM, Brunzell JD, Motulsky AG, Austin MA. Lipoprotein and apolipoprotein abnormalities in familial combined hyperlipidemia: a 20-year prospective study. Atherosclerosis. 2001 Dec;159(2):471-81. doi: 10.1016/s0021-9150(01)00528-7. PMID 11730829
- [Background] Carr MC, Hokanson JE, Zambon A, Deeb SS, Barrett PH, Purnell JQ, Brunzell JD. The contribution of intraabdominal fat to gender differences in hepatic lipase activity and low/high density lipoprotein heterogeneity. J Clin Endocrinol Metab. 2001 Jun;86(6):2831-7. doi: 10.1210/jcem.86.6.7586. PMID 11397895
- [Background] Carr MC, Brunzell JD. Abdominal obesity and dyslipidemia in the metabolic syndrome: importance of type 2 diabetes and familial combined hyperlipidemia in coronary artery disease risk. J Clin Endocrinol Metab. 2004 Jun;89(6):2601-7. doi: 10.1210/jc.2004-0432. PMID 15181030
- [Background] Brunzell JD, Iverius PH, Scheibel MS, Fujimoto WY, Hayden MR, McLeod R, Frolich J. Primary lipoprotein lipase deficiency. Adv Exp Med Biol. 1986;201:227-39. doi: 10.1007/978-1-4684-1262-8_20. PMID 3541517
- [Background] Brunzell JD, Fujimoto WY. Body fat distribution and dyslipidemia. Am J Med. 1995 Nov;99(5):457-8. doi: 10.1016/s0002-9343(99)80219-8. No abstract available. PMID 7485200